CLINICAL TRIAL: NCT06925555
Title: A Multi-center，Single-arm, Open-label Phase II Clinical Study on Brentuximab Vedotin Combined With Rituximab Plus Cyclophosphamide, Doxorubicin, and Prednisone (R-CHP) in the Treatment of Newly Diagnosed EBV-positive Diffuse Large B-cell Lymphoma, Not Otherwise Specified (EBV+ DLBCL-NOS)
Brief Title: Brentuximab Vedotin Combined With R-CHP in Newly Diagnosed EBV+ DLBCL-NOS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, M.D, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-050
Record Dates: First submitted 2025-04-10; First posted 2025-04-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: EBV-Positive Diffuse Large B-Cell Lymphoma, Nos; Brentuximab Vedotin
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BV+R-CHP Arm (Experimental): Newly Diagnosed EBV+ DLBCL-NOS Patients Receiving Brentuximab Vedotin plus R-CHP(Rituximab、Cyclophosphamide、Doxorubicin and Prednisone)
  Interventions: Drug: BV+R-CHP

INTERVENTIONS:
Drug: BV+R-CHP — Brentuximab Vedotin, 1.8mg/kg/dose, d0、Rituximab, 375 mg/m2, d0、Cyclophosphamide, 750 mg/m2, d1、Doxorubicin, 50 mg/m2, d1、Prednisone, 60mg/m2, d1-5

SUMMARY:
Evaluation of the Safety and Efficacy of Brentuximab Vedotin Combined With R-CHP in Newly Diagnosed EBV+ DLBCL-NOS.

DETAILED DESCRIPTION:
EBV-positive diffuse large B-cell lymphoma, not otherwise specified (EBV+ DLBCL-NOS), is an EBV-positive clonal B-cell lymphoid proliferation and circulating EBV-DNA is a great indicator for prognosis among EBV associated disease.Currently, there is no internationally standardized treatment regimen for EBV+DLBCL, NOS. There is an urgent clinical need to explore novel effective therapeutic strategies to improve survival in this patient population.CD30 is highly expressed in EBV+DLBCL, and CD30 positivity serves as an adverse prognostic factor.

Brentuximab Vedotin (BV), a CD30-targeted antibody-drug conjugate (ADC), has shown significant improvements in progression-free survival (PFS), overall survival (OS), and overall response rate (ORR) compared to placebo + lenalidomide + rituximab in relapsed/refractory DLBCL patients according to the ECHELON-3 study.Therefore, we propose a randomized, prospective, multicenter phase II clinical trial to evaluate the efficacy (PFS, ORR [CR/CRu + PR], CRR, OS) and safety profile of Brentuximab Vedotin combined with R-CHP (Rituximab, Cyclophosphamide, Doxorubicin,Prednisone) in newly diagnosed EBV+DLBCL, NOS patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients must meet all of the following inclusion criteria to be eligible for enrollment:

1. BV+DLBCL, NOS diagnosed by pathological diagnosis according to WHO 2016 classification criteria;
2. Sign the informed consent form;
3. Systemic PET/CT performed within 28 days prior to enrollment demonstrating at least one measurable lesion in two perpendicular dimensions (nodal lesion: longest diameter >15 mm, short axis >5 mm; extranodal lesion: longest diameter >10 mm) per Lugano 2014 criteria;
4. ECOG Performance Status (PS) of 0-2;
5. Adequate organ and bone marrow function defined as:

   * Hematology: Absolute neutrophil count (ANC) ≥1.0×10⁹/L, platelet count (PLT) ≥50×10⁹/L, hemoglobin (HGB) ≥8.0 g/dL; without granulocyte colony-stimulating factor, platelet transfusion, or red blood cell transfusion within 7 days prior to testing.
   * Liver function: Total bilirubin (TBIL) ≤1.5×ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN.
   * Renal function: Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance rate (CCR) ≥50 mL/min.
   * Cardiac function: NYHA class <III; left ventricular ejection fraction (LVEF) ≥50% by echocardiography.
   * Coagulation: International normalized ratio (INR) ≤1.5×ULN, activated partial thromboplastin time (APTT) ≤ULN +10 s, prothrombin time (PT) ≤ULN +3 s.
   * Thyroid function: Baseline thyroid-stimulating hormone (TSH) within normal range or abnormal TSH with normal T3/T4 levels and no clinical symptoms.
6. Expected survival ≥ 3 months.
7. Age 18-70 years.
8. For subjects of childbearing potential or with partners of childbearing potential: Agreement to use highly effective contraception during treatment and for 90 days after the last dose.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from the study：

  1. Central nervous system (CNS) involvement.
  2. Second primary malignancy (except cured non-melanoma skin cancer, superficial bladder cancer, cervical carcinoma in situ, gastrointestinal intramucosal carcinoma, or breast cancer with no recurrence within 5 years).
  3. History of severe allergic diseases, hypersensitivity to macromolecular protein preparations, or any component of Brentuximab Vedotin.
  4. Prior allogeneic organ transplant or hematopoietic stem cell transplantation.
  5. Concurrent systemic anti-tumor therapy during the study.
  6. Anti-cancer vaccines or immunostimulatory anti-tumor therapy within 3 months prior to enrollment.
  7. Active severe acute/chronic infection requiring systemic therapy.
  8. Active or history of autoimmune disease within 2 years (exceptions: vitiligo, psoriasis, alopecia, Graves' disease without systemic treatment in the past 2 years; hypothyroidism requiring thyroid hormone replacement only; type I diabetes controlled with insulin).
  9. Systemic immunosuppressive therapy within 4 weeks prior to enrollment (excluding topical/nasal/inhaled corticosteroids or physiologic doses ≤10 mg/day prednisone equivalent).
  10. Positive serology for HIV antibody (HIV-Ab), Treponema pallidum antibody (TP-Ab), HCV antibody (HCV-Ab); HBsAg-positive with HBV DNA >ULN.
  11. History of idiopathic pulmonary fibrosis or interstitial pneumonia.
  12. Active tuberculosis.
  13. Prior ≥Grade 3 immune-related adverse events from immunotherapy.
  14. History of neurologic/psychiatric disorders (e.g., epilepsy, dementia).
  15. Administration of live vaccines (e.g., influenza, varicella) within 4 weeks prior to treatment or planned during the study.
  16. History of alcohol/drug abuse.
  17. Pregnancy or lactation.
  18. Participation in another interventional clinical trial within 1 month prior to enrollment.
  19. Other factors deemed by investigators to potentially compromise efficacy/safety assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) rate | 2 years
  PFS was defined as the time between inclusion and the first date of progression, relapse, or death from any cause.

SECONDARY OUTCOMES:
ORR | every 3 cycles, up to 6 cycles (each cycle is 21 days)
  The Overall Response Rate
CR rate | every 3 cycles, up to 6 cycles (each cycle is 21 days)
  complete remission rate
2-year overall survival (OS) rate | 2 years
  Overall Survival: from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No